CLINICAL TRIAL: NCT03675126
Title: An Open-Label Extension Study for Patients With Duchenne Muscular Dystrophy Who Participated in Studies of SRP-5051
Brief Title: An Open-Label Extension Study for Patients With Duchenne Muscular Dystrophy Who Participated in Studies of SRP-5051 (Vesleteplirsen)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The sponsor has decided to integrate 5051-102 into 5051-201. Participants from 5051-102 will be eligible to enroll in 5051-201 Part B.
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5051-102
Record Dates: First submitted 2018-08-06; First posted 2018-09-18 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Muscular Dystrophy, Duchenne
Keywords: Duchenne muscular dystrophy; Exon Skipping; DMD; Exon 51; Ambulatory; Pediatric; Nonambulatory; Peptide-conjugated phosphorodiamidate morpholino oligomer (PPMO); Duchenne
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SRP-5051 (Experimental): Participants will receive SRP-5051 via intravenous (IV) infusion. Dosage and frequency will be determined from the safety profile of other ongoing SRP-5051 studies.
  Interventions: Drug: SRP-5051

INTERVENTIONS:
Drug: SRP-5051 — SRP-5051 administered as an IV infusion.
  Other Names: vesleteplirsen

SUMMARY:
The purpose of this extension study is to evaluate the safety, tolerability, and pharmacokinetics of repeat administrations of SRP-5051 (vesleteplirsen) in participants with Duchenne muscular dystrophy (DMD) who participated in studies of SRP-5051.

ELIGIBILITY:
Inclusion Criteria:

• Has completed a study of SRP-5051 and continues to meet the Eligibility Criteria of Study 5051-102.

Exclusion Criteria:

* Initiation or change of dosing (except for modifications to accommodate changes in weight or changes in standard of care) since completing a study administering SRP-5051 and while participating in this study for any of the following: angiotensin converting enzyme (ACE) inhibitors, angiotensin receptor blocking agents (ARBs), beta-blockers, potassium and steroids*.
* Requires antiarrhythmic and/or diuretic therapy for heart failure.
* Use of any herbal medication/supplement containing aristolochic acid.
* Treatment with any experimental therapy since entering original study or any experimental gene therapy for the treatment of DMD at any time.
* Participation in an interventional clinical trial since completing original study.

Other inclusion/exclusion criteria apply.

* The dose of steroids must remain constant except for modifications to accommodate changes in weight.

Min Age: 4 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2021-08-25 (Actual); Study Completion 2021-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sarepta Therapeutics, Inc.
Locations (8):
- United States (7):
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - NW FL Clinical Research Group, LLC, Gulf Breeze, Florida
  - Center for Integrative Rare Disease Research (CIRDR), Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Children's Medical Center Dallas, Dallas, Texas
- London Health Sciences Centre, London, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- SRP-5051: Participants received SRP-5051 via intravenous (IV) infusion every 4 weeks (Q4W).
Period: Overall Study
Arm/Group | SRP-5051
Started | 15
Received at Least 1 Dose of Study Drug | 15
Completed | 0
Not Completed | 15
Not completed — Study Terminated by Sponsor | 9
Not completed — Death | 2
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Population: Safety Set: all participants who started the study drug infusion.
Groups:
- SRP-5051: Participants received SRP-5051 via IV infusion Q4W.
Arm/Group | SRP-5051
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.5 (2.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 9
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs)
Description: A TEAE was any untoward medical occurrence in a clinical study participant that did not necessarily have a causal relationship with the study drug. A TEAE could, therefore, be any unfavorable and unintended symptom, sign, disease, condition, or test abnormality that occurred during or after administration of the study drug, whether or not considered related to the study drug. A summary of serious and all other non-serious TEAEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Up to approximately 135 weeks
Population: Safety Set: all participants who started the study drug infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | SRP-5051
Number analyzed (Participants) | 15
Participants | 14

2. Secondary Outcome: Plasma Concentration of SRP-5051
Description: For pharmacokinetic (PK) analysis, plasma samples were collected pre-dose (approximately 30 minutes prior to the start of infusion), immediately prior to the end of infusion (prior to flush), and approximately 4 to 6 hours after the end of dosing. Results are reported in micrograms/liter (ug/L) and are presented as an average across the days specified in the time frame.
Time Frame: Day 1, Day 84, every 84 days after Day 84 (up to a maximum of approximately 135 weeks) (pre-dose, immediately prior to end of infusion, up to 4-6 hours post-dose)
Population: Pharmacokinetic Set: all participants who started the study drug infusion and had at least 1 PK concentration data collection.
Measure: Mean (Standard Deviation); unit: ug/L
Arm/Group | SRP-5051
Number analyzed (Participants) | 15
ug/L
  Pre-dose | 486.25 (7717.595)
  End of Infusion | 45244.93 (42639.411)
  4-6 Hours Post-dose | 2790.32 (10941.464)

ADVERSE EVENTS:
Time Frame: Up to approximately 135 weeks
Description: Reported safety data based upon the Safety Set: all participants who started the study drug infusion.
Arm/Group | SRP-5051
All-Cause Mortality (participants affected / at risk) | 2/15
Serious Adverse Events (participants affected / at risk) | 6/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SRP-5051 (N=15)
Anaemia (Blood and lymphatic system disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiogenic shock (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Psychogenic seizure (Nervous system disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SRP-5051 (N=15)
Anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Atrioventricular block second degree (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Mucous stools (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 2
Catheter site pain (General disorders) | 1
Chest pain (General disorders) | 1
Injection site reaction (General disorders) | 1
Malaise (General disorders) | 1
Oedema peripheral (General disorders) | 1
Vessel puncture site bruise (General disorders) | 1
Bronchitis (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Tinea pedis (Infections and infestations) | 1
Tinea versicolour (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Contusion (Injury, poisoning and procedural complications) | 3
Fall (Injury, poisoning and procedural complications) | 3
Back injury (Injury, poisoning and procedural complications) | 1
Head injury (Injury, poisoning and procedural complications) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1
C-reactive protein increased (Investigations) | 2
Blood glucose increased (Investigations) | 1
Cystatin C increased (Investigations) | 1
Glucose urine present (Investigations) | 1
Total complement activity increased (Investigations) | 1
Troponin I increased (Investigations) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 7
Hypokalaemia (Metabolism and nutrition disorders) | 2
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Coccydynia (Musculoskeletal and connective tissue disorders) | 1
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 2
Dizziness postural (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 2
Crystalluria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Ketonuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1
Restrictive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Livedo reticularis (Skin and subcutaneous tissue disorders) | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Flushing (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Poor venous access (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/26/NCT03675126/Prot_000.pdf